CLINICAL TRIAL: NCT03979196
Title: Inpatient vs Outpatient Management of Women With Short Cervix: A Randomized Controlled Trial (RCT)
Brief Title: Inpatient vs Outpatient Management of Short Cervix
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Logistical Challenges
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: North York General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ShortCxTrial
Record Dates: First submitted 2019-06-05; First posted 2019-06-07 (Actual); Last update posted 2024-04-22 (Actual); Status verified 2024-04

CONDITIONS: Preterm Birth; Pregnancy, High Risk
Keywords: Preterm Birth; Pregnancy, High Risk; Short Cervix
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Inpatient Management (Active Comparator): Women in this arm will follow the standard of care for admission to high-risk units at Sunnybrook Health Sciences Centre or North York General Hospital.
  Interventions: Other: Inpatient Management
- Outpatient Management (Active Comparator): Women in this arm will be encouraged to follow the standard of care established in the high-risk clinics at Sunnybrook Health Sciences Centre or North York General Hospital.
  Interventions: Other: Outpatient Management

INTERVENTIONS:
Other: Inpatient Management — Admission for a minimum of three days, administration of betamethasone, and clinical reassessment by obstetrician after three days. After the initial three day admission, further management will be at the discretion of their obstetrician who will continue their care and decide if further admissions are needed.
  Weekly cervical length assessment will be performed until 28 weeks and patient readmission will be decided by their Obstetrician.
  Post-intervention, women in both arms will receive the same standard of care (weekly clinic or inpatient follow-up appointments) and will be followed to delivery. Prior to delivery, participants will complete a patient Quality of Life survey and at delivery, primary and secondary outcomes will be collected.
  Arms: Inpatient Management
Other: Outpatient Management — Avoid heavy lifting and core exercise, avoid intercourse, weekly assessment of cervical length by ultrasound and administration of betamethasone. Patients will continue with outpatient management for the remainder of their pregnancy with no admission unless the patient develops contractions, PPROM, bleeding, or the cervix is dilated to ≥1cm.
  Post-intervention, women in both arms will receive the same standard of care (weekly clinic or inpatient follow-up appointments) and will be followed to delivery. Prior to delivery, participants will complete a patient Quality of Life survey and at delivery, primary and secondary outcomes will be collected.
  Arms: Outpatient Management

SUMMARY:
The presence of short cervix during pregnancy is a risk factor for preterm birth though in many cases women will eventually deliver at term or near term.

While there are proven treatments such as cerclage and progesterone that can improve pregnancy outcomes, many women are advised to limit their activity, are put on bed rest, or admitted to hospital for inpatient management. Presently, there is no evidence that hospital admission of women with short cervix is beneficial and prolongs the pregnancy.

The investigators propose to examine whether inpatient management results in comparable outcomes to outpatient management for women with short cervix.

DETAILED DESCRIPTION:
Preterm birth, defined as the birth of a baby at less than 37 weeks' gestation, is a significant burden to society that is on the rise. Although many risk factors contribute to preterm birth, a short cervix is a well-established risk factor.The most common management for short cervix in Canada is vaginal progesterone, cervical cerclage, and hospital admission. Evidence suggests that vaginal progesterone and cervical cerclage improve outcomes, but there is very limited research on hospital admission or its efficacy. Due to the increased risk of preterm birth associated with cervical length ≤15 mm, some patients are admitted to hospital for observation even though labour is not imminent. The role of inpatient versus outpatient management is unclear and has not been explored. Hospital admission or modified activity has not been shown to improve pregnancy outcomes however, due to the increased risk of preterm birth, many women with short cervix are admitted for inpatient management.

This project's objective is to examine whether inpatient or outpatient care results in similar pregnancy outcomes for women with short cervix.

This is a multi-centre, non-inferiority randomized controlled trial in women with a singleton pregnancy and isolated short cervix (SC) (≤1.5cm by transvaginal scan (TVS)) at 23-28 weeks at Sunnybrook Health Sciences Centre (SHSC) and North York General Hospital (NYGH), in Toronto, Ontario, Canada. The intervention involves randomizing women to either inpatient or outpatient management and examining whether gestational age at delivery in women with SC (≤1.5cm by TVS) is comparable between arms. The investigators hypothesize that there will be no difference in the preterm birth rate and gestational age at delivery between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* Singleton pregnancy between 23 weeks 0 days - 28 weeks 6 days gestational age
* SC (≤1.5cm) determined by TVS
* Vaginal progesterone treatment
* Cervical dilatation of ≤1cm
* Located within 45 minute drive from recruitment site (Sunnybrook Health Sciences Centre or North York General Hospital)

Exclusion Criteria:

* Multiple pregnancy
* Preterm premature rupture of membranes (PPROM), vaginal bleeding, infection, high blood pressure (defined as 140/90 mm Hg or higher)
* Regular uterine contractions or active labour
* Vaginal bleeding
* Cervical dilatation of >1cm
* Fetal anomalies

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2019-06-06 (Actual); Primary Completion 2020-03-30 (Actual); Study Completion 2021-09-07 (Actual)

PRIMARY OUTCOMES:
Gestational age at delivery | At delivery

SECONDARY OUTCOMES:
Betamethasone treatment | Before delivery
Magnesium sulphate treatment | Before 32 weeks gestation
Intrapartum complications | During delivery
  Any of the following: cord prolapse, postpartum hemorrhage, or fetal distress
Mode of delivery | At delivery
  One of: vaginal delivery, caesarean section, operative delivery
Patient Quality of Life | 1 week after randomization
  36-Item Short Form Health Survey: 36-item, self-administered survey takes 5 minutes and is designed to measure health on eight multi-item dimensions, including functional status, well-being, and overall evaluation of health.
Neonatal morbidity and mortality: composite measure | 1-28 days post-delivery
  A composite of the following: Early-onset sepsis/meningitis (culture proven within first 7 days of life), Significant Intraventricular hemorrhage (IVH) (Grade III/IV, hemorrhagic venous infarct), Periventricular leukomalacia (PVL), Respiratory distress syndrome (RDS) (requiring surfactant and ventilation), Need for high frequency oscillatory ventilation (HFO) on Day 1, Need for inhaled nitric oxide (iNO) on Day 1, Pneumothorax (requiring needle aspiration or chest tube drainage), Chronic lung disease (requiring oxygen at discharge/transfer or at corrected gestational age (CGA) 36 weeks), Death, retinopathy of prematurity(ROP) (>Stage 2), necrotizing enterocolitis (NEC) (finding of pneumatosis, portal vein gas or free peritoneal air on abdominal radiograph), patent ductus arteriosus (PDA) (presence of PDA diagnosed by echocardiography or clinical suspicion treated with medication or surgery)

CONTACTS AND LOCATIONS:
Overall Officials: Ori Nevo, MD, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (2):
- Canada (2):
  - North York General Hospital, Toronto, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Menon R. Preterm birth: a global burden on maternal and child health. Pathog Glob Health. 2012 Jul;106(3):139-40. doi: 10.1179/204777312X13462106637729. No abstract available. PMID 23265368
- [Background] Blencowe H, Lee AC, Cousens S, Bahalim A, Narwal R, Zhong N, Chou D, Say L, Modi N, Katz J, Vos T, Marlow N, Lawn JE. Preterm birth-associated neurodevelopmental impairment estimates at regional and global levels for 2010. Pediatr Res. 2013 Dec;74 Suppl 1(Suppl 1):17-34. doi: 10.1038/pr.2013.204. PMID 24366461
- [Background] Blencowe H, Cousens S, Oestergaard MZ, Chou D, Moller AB, Narwal R, Adler A, Vera Garcia C, Rohde S, Say L, Lawn JE. National, regional, and worldwide estimates of preterm birth rates in the year 2010 with time trends since 1990 for selected countries: a systematic analysis and implications. Lancet. 2012 Jun 9;379(9832):2162-72. doi: 10.1016/S0140-6736(12)60820-4. PMID 22682464
- [Background] Alexander GR, Kogan M, Bader D, Carlo W, Allen M, Mor J. US birth weight/gestational age-specific neonatal mortality: 1995-1997 rates for whites, hispanics, and blacks. Pediatrics. 2003 Jan;111(1):e61-6. doi: 10.1542/peds.111.1.e61. PMID 12509596
- [Background] Institute of Medicine (US) Committee on Understanding Premature Birth and Assuring Healthy Outcomes; Behrman RE, Butler AS, editors. Preterm Birth: Causes, Consequences, and Prevention. Washington (DC): National Academies Press (US); 2007. Available from http://www.ncbi.nlm.nih.gov/books/NBK11362/ PMID 20669423
- [Background] Lawn JE, Cousens S, Zupan J; Lancet Neonatal Survival Steering Team. 4 million neonatal deaths: when? Where? Why? Lancet. 2005 Mar 5-11;365(9462):891-900. doi: 10.1016/S0140-6736(05)71048-5. PMID 15752534
- [Background] McCormick MC. The contribution of low birth weight to infant mortality and childhood morbidity. N Engl J Med. 1985 Jan 10;312(2):82-90. doi: 10.1056/NEJM198501103120204. PMID 3880598
- [Background] Berkowitz GS, Papiernik E. Epidemiology of preterm birth. Epidemiol Rev. 1993;15(2):414-43. doi: 10.1093/oxfordjournals.epirev.a036128. No abstract available. PMID 8174665
- [Background] Iams JD, Goldenberg RL, Meis PJ, Mercer BM, Moawad A, Das A, Thom E, McNellis D, Copper RL, Johnson F, Roberts JM. The length of the cervix and the risk of spontaneous premature delivery. National Institute of Child Health and Human Development Maternal Fetal Medicine Unit Network. N Engl J Med. 1996 Feb 29;334(9):567-72. doi: 10.1056/NEJM199602293340904. PMID 8569824
- [Background] Berghella V, Kuhlman K, Weiner S, Texeira L, Wapner RJ. Cervical funneling: sonographic criteria predictive of preterm delivery. Ultrasound Obstet Gynecol. 1997 Sep;10(3):161-6. doi: 10.1046/j.1469-0705.1997.10030161.x. PMID 9339522
- [Background] Berghella V, Roman A, Daskalakis C, Ness A, Baxter JK. Gestational age at cervical length measurement and incidence of preterm birth. Obstet Gynecol. 2007 Aug;110(2 Pt 1):311-7. doi: 10.1097/01.AOG.0000270112.05025.1d. PMID 17666605
- [Background] Crane JM, Hutchens D. Transvaginal sonographic measurement of cervical length to predict preterm birth in asymptomatic women at increased risk: a systematic review. Ultrasound Obstet Gynecol. 2008 May;31(5):579-87. doi: 10.1002/uog.5323. PMID 18412093
- [Background] Goldenberg RL, Iams JD, Das A, Mercer BM, Meis PJ, Moawad AH, Miodovnik M, VanDorsten JP, Caritis SN, Thurnau GR, Dombrowski MP, Roberts JM, McNellis D. The Preterm Prediction Study: sequential cervical length and fetal fibronectin testing for the prediction of spontaneous preterm birth. National Institute of Child Health and Human Development Maternal-Fetal Medicine Units Network. Am J Obstet Gynecol. 2000 Mar;182(3):636-43. doi: 10.1067/mob.2000.104212. PMID 10739521
- [Background] Guzman ER, Walters C, Ananth CV, O'Reilly-Green C, Benito CW, Palermo A, Vintzileos AM. A comparison of sonographic cervical parameters in predicting spontaneous preterm birth in high-risk singleton gestations. Ultrasound Obstet Gynecol. 2001 Sep;18(3):204-10. doi: 10.1046/j.0960-7692.2001.00526.x. PMID 11555447
- [Background] Heath VC, Southall TR, Souka AP, Elisseou A, Nicolaides KH. Cervical length at 23 weeks of gestation: prediction of spontaneous preterm delivery. Ultrasound Obstet Gynecol. 1998 Nov;12(5):312-7. doi: 10.1046/j.1469-0705.1998.12050312.x. PMID 9819868
- [Background] Owen J. Evaluation of the cervix by ultrasound for the prediction of preterm birth. Clin Perinatol. 2003 Dec;30(4):735-55. doi: 10.1016/s0095-5108(03)00103-9. PMID 14714921
- [Background] Ozdemir I, Demirci F, Yucel O, Erkorkmaz U. Ultrasonographic cervical length measurement at 10-14 and 20-24 weeks gestation and the risk of preterm delivery. Eur J Obstet Gynecol Reprod Biol. 2007 Feb;130(2):176-9. doi: 10.1016/j.ejogrb.2006.03.021. Epub 2006 May 8. PMID 16682111
- [Background] Cicero S, Skentou C, Souka A, To MS, Nicolaides KH. Cervical length at 22-24 weeks of gestation: comparison of transvaginal and transperineal-translabial ultrasonography. Ultrasound Obstet Gynecol. 2001 Apr;17(4):335-40. doi: 10.1046/j.1469-0705.2001.00345.x. PMID 11339192
- [Background] Yazici G, Yildiz A, Tiras MB, Arslan M, Kanik A, Oz U. Comparison of transperineal and transvaginal sonography in predicting preterm delivery. J Clin Ultrasound. 2004 Jun;32(5):225-30. doi: 10.1002/jcu.20027. PMID 15124188
- [Background] Andersen HF, Nugent CE, Wanty SD, Hayashi RH. Prediction of risk for preterm delivery by ultrasonographic measurement of cervical length. Am J Obstet Gynecol. 1990 Sep;163(3):859-67. doi: 10.1016/0002-9378(90)91084-p. PMID 2206073
- [Background] Hassan SS, Romero R, Vidyadhari D, Fusey S, Baxter JK, Khandelwal M, Vijayaraghavan J, Trivedi Y, Soma-Pillay P, Sambarey P, Dayal A, Potapov V, O'Brien J, Astakhov V, Yuzko O, Kinzler W, Dattel B, Sehdev H, Mazheika L, Manchulenko D, Gervasi MT, Sullivan L, Conde-Agudelo A, Phillips JA, Creasy GW; PREGNANT Trial. Vaginal progesterone reduces the rate of preterm birth in women with a sonographic short cervix: a multicenter, randomized, double-blind, placebo-controlled trial. Ultrasound Obstet Gynecol. 2011 Jul;38(1):18-31. doi: 10.1002/uog.9017. Epub 2011 Jun 15. PMID 21472815
- [Background] Jarde A, Lutsiv O, Park CK, Beyene J, Dodd JM, Barrett J, Shah PS, Cook JL, Saito S, Biringer AB, Sabatino L, Giglia L, Han Z, Staub K, Mundle W, Chamberlain J, McDonald SD. Effectiveness of progesterone, cerclage and pessary for preventing preterm birth in singleton pregnancies: a systematic review and network meta-analysis. BJOG. 2017 Jul;124(8):1176-1189. doi: 10.1111/1471-0528.14624. Epub 2017 Apr 17. PMID 28276151
- [Background] Sotiriadis A, Papatheodorou S, Kavvadias A, Makrydimas G. Transvaginal cervical length measurement for prediction of preterm birth in women with threatened preterm labor: a meta-analysis. Ultrasound Obstet Gynecol. 2010 Jan;35(1):54-64. doi: 10.1002/uog.7457. PMID 20014326
- [Background] Sosa C, Althabe F, Belizan J, Bergel E. Bed rest in singleton pregnancies for preventing preterm birth. Cochrane Database Syst Rev. 2004;(1):CD003581. doi: 10.1002/14651858.CD003581.pub2. PMID 14974024
- [Background] Fox NS, Jean-Pierre C, Predanic M, Chasen ST. Does hospitalization prevent preterm delivery in the patient with a short cervix? Am J Perinatol. 2007 Jan;24(1):49-53. doi: 10.1055/s-2006-958164. Epub 2006 Dec 27. PMID 17195150
- [Background] Grobman WA, Gilbert SA, Iams JD, Spong CY, Saade G, Mercer BM, Tita ATN, Rouse DJ, Sorokin Y, Leveno KJ, Tolosa JE, Thorp JM, Caritis SN, Peter Van Dorsten J; Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) Maternal-Fetal Medicine Units (MFMU) Network*. Activity restriction among women with a short cervix. Obstet Gynecol. 2013 Jun;121(6):1181-1186. doi: 10.1097/AOG.0b013e3182917529. PMID 23812450
- [Background] Shea AK, Simpson AN, Barrett J, Ladhani N, Nevo O. Pregnancy Outcomes of Women Admitted to a Tertiary Care Centre with Short Cervix. J Obstet Gynaecol Can. 2017 May;39(5):328-334. doi: 10.1016/j.jogc.2017.01.012. PMID 28454755
- [Background] Ware JE Jr, Sherbourne CD. The MOS 36-item short-form health survey (SF-36). I. Conceptual framework and item selection. Med Care. 1992 Jun;30(6):473-83. PMID 1593914
- [Background] Provencher et al. Fertility: Overview, 2012 to 2016. Reports on the Demographic Situation in Canada. 2018; Catalogue no. 91-209-X.
- [Background] Copyright © 2013, SAS Institute Inc., Cary, NC, USA.